CLINICAL TRIAL: NCT00554905
Title: Radiofrequency Ablation With or With Transcatheter Arterial Embolization for Hepatocellular Carcinoma
Acronym: RFA and TACE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Cancer Center, Sun Yat-sen University, Cancer Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rfa-001
Record Dates: First submitted 2007-11-06; First posted 2007-11-07 (Estimated); Last update posted 2009-02-10 (Estimated); Status verified 2009-02

CONDITIONS: Hepatocellular Carcinoma; Liver Cancer
Keywords: ablation; catheter; Carcinoma, Hepatocellular; therapy; Chemoembolization, Therapeutic; Humans; Liver Neoplasms
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): TACE first, then RFA within 2 weeks
  Interventions: Procedure: Radiofrequency ablation; Procedure: TACE
- 2 (Active Comparator): RFA alone
  Interventions: Procedure: Radiofrequency ablation

INTERVENTIONS:
Procedure: Radiofrequency ablation — For RFA, we used a commercially available system (RF 2000; Radio Therapeutics, Mountain View, California, USA) and a needle electrode with a 15-gauge insulated cannula with 10 hook-shape expandable electrode tines with a diameter of 3.5cm at expansion (LeVeen; RadioTherapeutics, Mountain View, California, USA).
  Other Names: RFA
Procedure: TACE — TACE first, then RFA within 2 weeks
  Other Names: RFA-TACE
  Arms: 1

SUMMARY:
The purpose of this study is to prospectively evaluate whether combined RFA and TACE (RFA-TACE) result in better survival outcomes than RFA alone in patients with HCC.

DETAILED DESCRIPTION:
Local ablation is a safe and effective therapy for patients who cannot undergo resection, or as a bridge to transplantation. Of the various percutaneous local ablative therapies, radiofrequency ablation (RFA) has attracted the greatest interest because of its effectiveness and safety for small HCC ≤ 5.0cm, with a 3-year survival rate of 62% to 68%, a low treatment morbidity of 0% to 12%, and a low treatment mortality of 0% to 1%. Prospective randomized trials have shown RFA to be better than percutaneous ethanol injection (PEI) in producing a higher rate of complete tumor necrosis with fewer numbers of treatment sessions and better survival.

Unfortunately, the complete tumor necrosis rate for tumors larger than 5cm is less favorable, and the local recurrence rate can be as high as 20% even in small HCC less than 3.5cm. The high local recurrence rate may be due to residual cancer cells not killed by RFA or adjacent microscopic satellite tumor nodules.

Transcatheter Arterial Chemoembolization (TACE) is proved to be an effective and palliative therapy for unresectable HCC. And some studies showed that combined TACE and RFA may produce superior tumor control than RFA alone and reduce local recurrence rate. In a study by Yamakado et al., 64 patients with 92 tumors underwent RFA within two weeks after TACE. The intrahepatic recurrence rates were 15% at 1 year and 43% at 2years, the 1, and 2, year overall survivals were 100% and 93%, respectively. These results appeared favorable, but there has not a prospective randomized controlled study to compare RFA combine with TACE versus RFA alone.

Thus the purpose of our study was to prospectively evaluate whether combined RFA and TACE (RFA-TACE) result in better survival outcomes than RFA alone in patients with HCC.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 75 years, who refused surgery
* A solitary HCC ≤ 7.0cm in diameter, or multiple HCC ≤ 3 lesions, each ≤ 3.0cm in diameter
* Lesions being visible on ultrasound (US) and with an acceptable/safe path between the lesion and the skin as shown on US
* No extrahepatic metastasis
* No imaging evidence of invasion into the major portal/hepatic vein branches
* No history of encephalopathy, ascites refractory to diuretics or variceal bleeding
* A platelet count of > 40,000/mm3
* No previous treatment of HCC except liver resection

Exclusion Criteria:

* Patient compliance is poor
* The blood supply of tumor lesions is absolutely poor or arterial-venous shunt that TACE can not be performed
* Previous or concurrent cancer that is distinct in primary site or histology from HCC, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis & T1). Any cancer curatively treated > 3 years prior to entry is permitted.
* History of cardiac disease:

  * Congestive heart failure > New York Heart Association (NYHA) class 2
  * Active coronary artery disease (myocardial infarction more than 6 months prior to study entry is permitted)
  * Cardiac arrhythmias requiring anti-arrhythmic therapy other than beta blockers, calcium channel blocker or digoxin; or
  * Uncontrolled hypertension (failure of diastolic blood pressure to fall below 90 mmHg, despite the use of 3 antihypertensive drugs).
* Active clinically serious infections (> grade 2 National Cancer Institute [NCI]-Common Terminology Criteria for Adverse Events [CTCAE] version 3.0)
* Known history of human immunodeficiency virus (HIV) infection
* Known central nervous system tumors including metastatic brain disease
* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry
* Distantly extrahepatic metastasis
* History of organ allograft
* Substance abuse, medical, psychological or social conditions that may interfere with the patient's participation in the study or evaluation of the study results
* Known or suspected allergy to the investigational agent or any agent given in association with this trial
* Any condition that is unstable or which could jeopardize the safety of the patient and his/her compliance in the study
* Pregnant or breast-feeding patients. Women of childbearing potential must have a negative pregnancy test performed within seven days prior to the start of study drug. Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial.
* Excluded therapies and medications, previous and concomitant:

  * Prior use of any systemic anti-cancer treatment for HCC, eg. chemotherapy, immunotherapy or hormonal therapy (except that hormonal therapy for supportive care is permitted). Antiviral treatment is allowed, however interferon therapy must be stopped at least 4 weeks prior randomization.
  * Prior use of systemic investigational agents for HCC
  * Autologous bone marrow transplant or stem cell rescue within four months of start of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2006-10; Primary Completion 2009-02 (Estimated); Study Completion 2009-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 3, 5 years

SECONDARY OUTCOMES:
Recurrence rates | 3, 5-years

CONTACTS AND LOCATIONS:
Overall Officials: Min-Shan Chen, Doctor, Principal Investigator — Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University; Jin-Qing Li, Doctor, Study Chair — Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University
Locations (1):
- Department of Hepatobilliary Surgery, Cancer Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Bruix J, Sherman M; Practice Guidelines Committee, American Association for the Study of Liver Diseases. Management of hepatocellular carcinoma. Hepatology. 2005 Nov;42(5):1208-36. doi: 10.1002/hep.20933. No abstract available. PMID 16250051
- [Derived] Peng ZW, Zhang YJ, Chen MS, Xu L, Liang HH, Lin XJ, Guo RP, Zhang YQ, Lau WY. Radiofrequency ablation with or without transcatheter arterial chemoembolization in the treatment of hepatocellular carcinoma: a prospective randomized trial. J Clin Oncol. 2013 Feb 1;31(4):426-32. doi: 10.1200/JCO.2012.42.9936. Epub 2012 Dec 26. PMID 23269991